CLINICAL TRIAL: NCT07117890
Title: a Study of Sunvozertinib Treatment in Untreated Advanced NSCLC With EGFR Uncommon Mutations
Brief Title: Sunvozertinib Treatment in Untreated Advanced NSCLC With EGFR Uncommon Mutations
Acronym: WU-KONG35
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Chief physician, Fudan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUM-NSCLC-01
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Sunvozertinib; EGFR; EGFR uncommon mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunvozertinib 300mg (Experimental): sunvozertinib monotherapy, 300mg QD
  Interventions: Drug: sunvozertinib 300mg
- sunvozertinib 200mg (Experimental): sunvozertinib monotherapy, 200mg QD
  Interventions: Drug: sunvozertinib 200mg

INTERVENTIONS:
Drug: sunvozertinib 300mg — sunvozertinib monotherapy, 300mg QD
  Arms: Sunvozertinib 300mg
Drug: sunvozertinib 200mg — sunvozertinib monotherapy, 200mg QD
  Arms: sunvozertinib 200mg

SUMMARY:
This study is a single arm study to access the anti-tumor efficacy and safety of sunvozertinib in untreated advanced NSCLC patients with EGFR uncommon mutations.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. histologically or cytologically confirmed non-squamous NSCLC with documented EGFR uncommon mutations from a local laoratory. at least one EGFR uncommon mutation (excluding EGFR 19del/l858r/T790m/Ex 20ins ) or compund mutations with EGFR uncommon mutations.
3. predicted life expectancy ≥ 12 weeks.
4. patient must have measurable disease according to RECIST 1.1

Exclusion Criteria:

1. previos systemic anti-tumor therapy
2. a history of malignant tumors within 2years
3. any severa or poorly controlled systemic disease per investigator's judgement
4. active infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | from first dose to last dose ,up to 24 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) | from first dose to first documented disease progression assessed by investigator or death due to any cause up to 48 months ,up to 18 months
Duration of Response (DoR) | for subject with PR or CR defined as the time from the first dose documentd CR or PR to disease progression or death up to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan university shanghai cancer center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No